CLINICAL TRIAL: NCT03455114
Title: A Single-arm, Open-label Feasibility Study for Assessing the Safety and Performance of the Modified AssiAnchor
Acronym: cataracts
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hanita Lenses (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AssiAnchor-02
Record Dates: First submitted 2018-02-11; First posted 2018-03-06 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- capsular fixation surgery (Experimental): patients required capsule centration safely undergo capsular fixation surgery with AssiAnchor under local anesthesia .
  Interventions: Device: AssiAnchor

INTERVENTIONS:
Device: AssiAnchor — The novel device, the capsular "Anchor", was designed to secure the capsular bag to the scleral wall. The device is a one-piece, one-plane intraocular implant . It works like a paper clip; holding the anterior capsule between a central rod, placed in front of the capsule, and the two lateral arms, inserted through the eye surgery and placed behind the capsule.

SUMMARY:
The AssiAnchor 2 is a fixation ophthalmic device. The device is manufactured by Hanita Lenses from PMMA material which is being used for the production of Intra-ocular lenses.

The device is intended for patients requiring capsule centration to clip the anterior lens capsule between the arms of the device and secure it to the scleral wall.

DETAILED DESCRIPTION:
Intended Use:

The AssiAnchor is a device which is intended to be implanted permanently in the posterior chamber of the eye for fixation of subluxated capsule.

Study Objectives:

The primary aim of this study is to assess the safety and performance of the new AssiAnchor. Safety will be assessed by evaluating the rate of adverse events and adverse device effects occurred throughout the study period.

Study population:

Men and women diagnosed with subluxated capsular bag that require lens removal surgery or in malpositioned pseudophakia that meet the inclusion/exclusion criteria and provide written informed consent will be enrolled in the study.

Enrollment:

A total of 10 subjects will be enrolled.

Investigational sites:

One (1) center will participate in this study.

Duration of Subject participation:

Completion of active enrolment is anticipated to last approximately 12 months. The objectives of this study will be achieved when the final study subject has completed 3 months follow-up.

Primary Safety Endpoint :

* Ease of implantation.
* Stability of device within the eye

Secondary Performance Endpoints -:

IOL stability, centration and tilt, visual acuity

Study Group:

A single study group. This is a single arm design; there is no control device in this study.

Key Inclusion Criteria:

Subject requires capsule centration. Subject is between 18 and 100 years of age Subject understands the study requirements and the treatment procedures and provides written Informed Consent before any study-specific tests or procedures are performed

Key Exclusion Criteria:

Subject is diagnosed with active anterior segment intraocular inflammation Subject is obligated to previous participation in another study with any investigational drug or device within the past 30 days Subject is pregnant

Visits & Procedures Pre-operative visit: 0-1 month prior the implantation procedure. The visit will include subject's qualification assessment for inclusion/exclusion criteria as described above. Informed consent must be signed.

Complete anamnesis will be taken including subject's medical complaints, medical history, medication use and ophthalmic examinations, family history and any detail relevant to the cause of lens malposition Surgical procedure: Procedure will be performed under anesthesia (at physician discretion) and the modified AssiAnchor will be implanted.

Follow-up: All subjects will have regularly follow-up visits up to 3 months post-implantation. All postoperative visits will include a complete ophthalmic examinations, medications used and recording of adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Requires capsule centration during or after cataract surgery.
* Understands the study requirements and the treatment procedures
* Sign Informed Consent before any study-specific tests or procedures.

Exclusion Criteria:

* Diagnosed with active anterior segment intraocular inflammation.
* Obligated to participation in another clinical study within the past 30 days.
* Pregnant.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-03-24 (Actual); Primary Completion 2021-06-09 (Actual); Study Completion 2021-06-09 (Actual)

PRIMARY OUTCOMES:
Safety of the new AssiAnchor. | 1 year
  Stability of device with in the eye will be assessed
performance of the new AssiAnchor. | 1 year
  We will assess if implantation of AssiAnchor
  * Enables cataract surgery for subluxated lens
  * Centers subluxated capsule
  * Provides a wide contact between the device and the anterior capsule

CONTACTS AND LOCATIONS:
Locations (1):
- MeirMC, Kfar Saba, Israel